CLINICAL TRIAL: NCT04780503
Title: The Rapid Shallow Breathing Index as an Early Predictor for Intubation and Mortality in Patients Undergoing Non-invasive Mechanical Ventilation in Acute Respiratory Failure
Brief Title: The Value of Rapid Shallow Breathing Indeks in Predicting Non-invasive Mechanical
Acronym: RSBI
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Emergency Medicine Specialist, Izmir Katip Celebi University
Other Study IDs: 2020-GOKAE-0011
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intubation Group/ Non-Intubation Group: Intubation group: Patients who failed noninvasive mechanical ventilation and who underwent endotracheal intubation Non-Intubation Group: Patients whose noninvasive mechanical ventilation is successful and endotracheal intubation is not applied
  Interventions: Diagnostic Test: Rapid Shallow Breathing Index
- Dying patients / Surviving patients: Dying patients :Patients with in-hospital mortality presenting with acute respiratory failure Surviving patients: Patients presenting and surviving due to acute respiratory failure
  Interventions: Diagnostic Test: Rapid Shallow Breathing Index

INTERVENTIONS:
Diagnostic Test: Rapid Shallow Breathing Index — The RSBI is defined as the ratio of respiratory frequency to tidal volume.

SUMMARY:
There are some criteria such as the most frequently used parameters to predict the failure of non-invasive mechanical ventilation, the APACHE 2 score, the presence of pneumonia and ARDS in the etiology, and no improvement in one hour of treatment. However, APECHE 2 score, which is the broadest of these criteria and includes others, is a complex scoring in which a large number of parameters are evaluated together, dependent on laboratory results and still leaves the final decision to the physician with a complete evaluation. In addition, the APACHE 2 score is a more commonly used method for intensive care patients rather than emergency patients who need a quick decision. Therefore, there is a need for a fast and practical method that can predict NIMV failure and determine early intubation decision in the management of patients admitted to the emergency department with acute dyspnea. Rapid Shallow Breathing Index (RSBI) is a parameter calculated by dividing the respiratory rate by the tidal volume and is used to predict whether patients who are intubated in intensive care unit can be extubated successfully.

The aim of this study is to evaluate the success of RSBI in predicting intubation and mortality in patients presented to the emergency department with acute respiratory failure and had NIMV indication.

DETAILED DESCRIPTION:
Respiratory failure is a challenging health problem that constitutes a significant part of emergency room visits (1). Acute respiratory failure treatment is a complex process in which pharmacological and non-pharmacological methods are used in combination. Non-invasive Mechanical Ventilation (NIMV) and Invasive Mechanical Ventilation (IMV) are life-saving methods commonly used in the emergency department in severe respiratory failure (2). In patients with severe dyspnea, NIMV improves alveolar gas exchange, with very successful results in selected patients (3). However, while NIMV cannot be used in patients who are unconscious, unable to protect the airway, have upper gastrointestinal bleeding and facial trauma and cannot adapt to non-invasive mechanical ventilation, these patients have IMV indication. Both methods are quite successful when used in selected cases. Therefore, patient selection is very important for NIMV and IMV (4). It is known that endotracheal intubation increases the risk of developing complications such as ventilator-associated pneumonia and sepsis. Therefore, unnecessary endotracheal intubation and invasive mechanical ventilation therapy are expected to increase mortality (5). On the other hand, delayed intubation decision is known to be an independent risk factor for increased mortality when NIMV fails (6) (7) (8). A method that predicts NIMV failure and enables effective mortality estimation may be useful in facilitating patient selection and providing appropriate treatment to patients. There are some criteria predicting that NIMV will fail in patients with severe respiratory distress and may be guiding for early intubation. The most commonly used of these are high APACHE 2 score, ARDS or pneumonia as the etiology of respiratory distress, advanced age, and no clinical improvement after 1 hour of treatment (9). However, APECHE 2 score, which is the broadest of these criteria and includes others, is a complex scoring in which a large number of parameters are evaluated together, dependent on laboratory results and still leaves the final decision to the physician with a complete evaluation. In addition, the APACHE 2 score is a more commonly used method for intensive care patients rather than emergency patients who need a quick decision. Therefore, there is a need for a fast and practical method that can predict NIMV failure and determine early intubation decision in the management of patients admitted to the emergency department with acute dyspnea. Rapid Shallow Breathing Index (RSBI) is a parameter calculated by dividing the respiratory rate by the tidal volume and is used to predict whether patients who are intubated in intensive care unit can be extubated successfully (10). In a study by Berg et al. (11) evaluating the endotracheal intubation and mortality rates of patients who underwent NIMV, it was found that the RSBI value above 105 obtained with a single measurement was significant in predicting NIV failure. Although this result is significant, it is not sufficient to make an early intubation decision. Considering that serial measurements are found to be more meaningful than a single measurement while predicting weaning success (12), serial measurements can provide more successful results in predicting intubation and mortality of patients receiving NIMV. Although the RSBI value obtained immediately after the initiation of NIMV is high, it is possible for the patient to be relieved after the patient has been treated with NIMV for a while and thus, the RSBI value may also decrease. For this reason, after these patients have been treated for a while, obtaining RSBI value once again and looking at the patient's response to treatment may provide more meaningful results.

The aim of this study is to evaluate the success of RSBI in predicting intubation and mortality in patients presented to the emergency department with acute respiratory failure and had NIMV indication.

ELIGIBILITY:
Inclusion Criteria:

* This study included patients 18 years of age and older with acute respiratory failure of any etiology and in need of NIVM. NIMV Initiation Criteria;
* Presentation of acute respiratory acidosis (pH ⩽7.35)
* Tachypnea (respiratory rate >20-24 breaths/minute) despite the standart medical teraphy
* Arterial oxygen tension/inspiratory oxygen fraction ratio (PaO2/FIO2) ⩽200

Exclusion Criteria:

* Pregnancy, trauma, NIMV intolerance and IMV initiation criteria;
* Cardiac or respiratory arrest
* Unstable cardiac arrhythmias
* Hemodynamic instability
* Severe encephalopathy (GCS <10)
* Severe upper gastrointestinal bleeding
* Facial trauma
* Upper airway obstruction
* Inability to protect the airway

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of only patients (patients admitted to the emergency department with acute respiratory failure)
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Rapid Shallow Breathing Index (RSBI) | 0-30 minute.
  The RSBI is the ratio of respiratory frequency to tidal volume (f/VT). RSBI values measured at admission and 30 minutes are the primary outcome measures of the study.

SECONDARY OUTCOMES:
Mean arterial pressure | 0-30 minute
  It is obtained by summing twice the diastolic pressure with the systolic pressure and dividing the obtained value by 3.
Respiratory rate | 0-30 minute
  It refers to the patient's respiratory rate in 1 minute.
Heart rate | 0-30 minute
  It refers to the patient's Heart rate in 1 minute.
Oxygen saturation | 0-30 minute
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Topal, MD, Study Chair — Izmir Katip Celebi University
Locations (1):
- IKCU, Ataturk Training and Research Hospital, Department of Emergency Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We have a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Chatila W, Jacob B, Guaglionone D, Manthous CA. The unassisted respiratory rate-tidal volume ratio accurately predicts weaning outcome. Am J Med. 1996 Jul;101(1):61-7. doi: 10.1016/s0002-9343(96)00064-2. PMID 8686717
- [Result] Shrestha AP, Shrestha R, Shrestha SK, Pradhan A. Prevalence of Dyspnea among Patients Attending the Emergency Department of a Tertiary Care Hospital: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2019 Sep-Oct;57(219):302-306. doi: 10.31729/jnma.4582. PMID 32329452
- [Result] Huang CC, Muo CH, Wu TF, Chi TY, Shen TC, Hsia TC, Shih CM. The application of non-invasive and invasive mechanical ventilation in the first episode of acute respiratory failure. Intern Emerg Med. 2021 Jan;16(1):83-91. doi: 10.1007/s11739-020-02315-1. Epub 2020 Mar 30. PMID 32232782
- [Result] Mas A, Masip J. Noninvasive ventilation in acute respiratory failure. Int J Chron Obstruct Pulmon Dis. 2014 Aug 11;9:837-52. doi: 10.2147/COPD.S42664. eCollection 2014. PMID 25143721
- [Result] Hayzy RC, McSpasson JI. Noninvasive ventilation in adults with acute respiratory failure: Benefits and contraindications. In: UpToDate, Post, TW (Ed), UpToDate, Waltham, MA, 2020.
- [Result] Girou E, Schortgen F, Delclaux C, Brun-Buisson C, Blot F, Lefort Y, Lemaire F, Brochard L. Association of noninvasive ventilation with nosocomial infections and survival in critically ill patients. JAMA. 2000 Nov 8;284(18):2361-7. doi: 10.1001/jama.284.18.2361. PMID 11066187
- [Result] Esteban A, Frutos-Vivar F, Ferguson ND, Arabi Y, Apezteguia C, Gonzalez M, Epstein SK, Hill NS, Nava S, Soares MA, D'Empaire G, Alia I, Anzueto A. Noninvasive positive-pressure ventilation for respiratory failure after extubation. N Engl J Med. 2004 Jun 10;350(24):2452-60. doi: 10.1056/NEJMoa032736. PMID 15190137
- [Result] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Result] Demoule A, Chevret S, Carlucci A, Kouatchet A, Jaber S, Meziani F, Schmidt M, Schnell D, Clergue C, Aboab J, Rabbat A, Eon B, Guerin C, Georges H, Zuber B, Dellamonica J, Das V, Cousson J, Perez D, Brochard L, Azoulay E; oVNI Study Group; REVA Network (Research Network in Mechanical Ventilation). Changing use of noninvasive ventilation in critically ill patients: trends over 15 years in francophone countries. Intensive Care Med. 2016 Jan;42(1):82-92. doi: 10.1007/s00134-015-4087-4. Epub 2015 Oct 13. PMID 26464393
- [Result] Antonelli M, Conti G, Moro ML, Esquinas A, Gonzalez-Diaz G, Confalonieri M, Pelaia P, Principi T, Gregoretti C, Beltrame F, Pennisi MA, Arcangeli A, Proietti R, Passariello M, Meduri GU. Predictors of failure of noninvasive positive pressure ventilation in patients with acute hypoxemic respiratory failure: a multi-center study. Intensive Care Med. 2001 Nov;27(11):1718-28. doi: 10.1007/s00134-001-1114-4. Epub 2001 Oct 16. PMID 11810114
- [Result] Karthika M, Al Enezi FA, Pillai LV, Arabi YM. Rapid shallow breathing index. Ann Thorac Med. 2016 Jul-Sep;11(3):167-76. doi: 10.4103/1817-1737.176876. PMID 27512505
- [Result] Berg KM, Lang GR, Salciccioli JD, Bak E, Cocchi MN, Gautam S, Donnino MW. The rapid shallow breathing index as a predictor of failure of noninvasive ventilation for patients with acute respiratory failure. Respir Care. 2012 Oct;57(10):1548-54. doi: 10.4187/respcare.01597. Epub 2012 Mar 12. PMID 22417884